CLINICAL TRIAL: NCT02323139
Title: A Single-arm Dose Finding Phase Ib Multicenter Study of the Oral Smoothened Antagonist LDE255 in Combination With Azacitidine for High Risk Myelodysplastic Syndrome Patients
Brief Title: A Study of LDE255 in Combination With Azacitidine for High Risk Myelodysplastic Syndrome Patients
Acronym: LDE255
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GFM-AZA-LDE; 2013-003108-38 (EudraCT Number)
Record Dates: First submitted 2014-05-26; First posted 2014-12-23 (Estimated); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: MDS
Keywords: High risk MDS; Azacitidine; LDE255
MeSH Terms: interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combination of azacitidine and LDE255 (Experimental): Combination of azacitidine at maximum tolerated dose and LDE255 at dose escalation, the starting dose will be 400 mg
  Interventions: Drug: Azacitidine and LDE255

INTERVENTIONS:
Drug: Azacitidine and LDE255 — Azacitidine at maximum tolerated dose. LDE255 at dose escalation (200, 400 or 800 mg)
  Other Names: Vidaza

SUMMARY:
This study is a phase Ib add-on study of the combination of LDE255 to azacitidine in patients without marrow response after at least 6 cycles of azacitidine.

DETAILED DESCRIPTION:
Dose escalation of LDE255 will be performed over time using a rolling 6 design to determine the safety of the combination with azacitidine. The starting dose will be 400 mg. Azacitidine will be continued at maximum tolerated dose (MTD). Evaluation will be based on cycle 1 toxicity profile. Once MTD will be determined, 20 additional patients will be treated at recommended dose.

ELIGIBILITY:
Inclusion Criteria:

1. High risk myelodysplastic syndrome (MDS) according to International Prognosis Scoring System (IPSS) or acute myeloid leukemia (AML) with low blast count (Bone marrow blast count between 20 and 30%) or non proliferative chronic myelomonocytic leukemia (CMML) (White blood cell (WBC) below 13 G/L)
2. Age over 18 years
3. Performance Status 0 to 2
4. Patient must have recovered from toxicities of any prior treatment regimen (no common toxicity criteria for adverse events (CTCAE)) grading over 1 for non-hematological toxicities, return to baseline for hematological values)
5. Patient must have been treated with azacitidine single agent for at least 6 cycles
6. According to International working group (IWG) 2006 criteria, patient may have a/ stable disease, OR b/ disease progression limited to patients with loss of hematological improvement without bone marrow progression. Patients with bone marrow progression (i.e. increased bone marrow blast count of 50% or more) should not be included.
7. Bone marrow blast count should be 10% to 30%
8. Adequate liver and renal function:

   * Serum creatinine less than 1.5 x the institutional upper limit of normal (ULN)
   * Total bilirubin less than 1.5 x the ULN unless considered due to Gilbert's syndrome
   * Alanine aminotransferase (ALT, SGPT), or aspartate aminotransferase (AST, SGOT) less than 2.5 x the ULN unless considered due to organ leukemic involvement
   * Creatine Kinase less than 1.5 x the ULN
9. Able to understand and sign the written informed consent
10. Women of childbearing potential must agree to use effective contraception without interruption throughout the study and for a further 3 months after the end of treatment
11. Men must agree to not conceive during the treatment and to use effective contraception during the treatment period (including periods of dose reduction or temporary suspension) and for a further 3 months after the end of treatment if their partner is of childbearing potential.

Exclusion Criteria:

1. Allogeneic stem cell transplantation (SCT) within the last 4 months and/or active graft versus host disease (GVHD), or autologous SCT within the last 4 weeks. Patient suitable for allogeneic transplantation and with an identified allogeneic donor (Extension phase only).
2. Active central nervous system (CNS) leukemic involvement.
3. Major surgery within 2 weeks of initiation of study medication.
4. Concurrent uncontrolled medical conditions that may interfere or potentially affect the interpretation of the study.
5. Unable to take oral drugs, or lack of physical integrity of the upper gastrointestinal tract, or known malabsorption syndromes.
6. Patients with unresolved diarrhea > CTCAE grade 2.
7. Patients who have previously been treated with systemic LDE225 or with other Hh pathway inhibitors.
8. Patients who have neuromuscular disorders (i.e. inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis and spinal muscular atrophy) or are on concomitant treatment with drugs that are recognized to cause rhabdomyolysis, such as 3-hydroxy-3-methylglutaryl-coenzyme A (HMG CoA) inhibitors (statins), clofibrate and gemfibrozil. Pravastatin may be used if necessary, with extra caution.
9. Patients who are planning on embarking on new physical activities, such as strenuous exercise, that can result in significant increases in plasma creatine kinase levels while on study treatment. Strenuous muscular activity MUST be avoided within 1 week of blood tests during the study.
10. Patient has history of cardiac dysfunction including any of the following:

    * Myocardial infarction documented by elevated cardiac enzymes or persistent regional wall abnormalities on assessment of life ventricular ejection fraction (LVEF) function within the last six months.
    * History of documented congestive heart failure (New York Association functional classification III-IV).
    * Documented cardiomyopathy.
    * Familial history of long QT syndrome.
11. Patient has active cardiac disease including any of the following:

    * Corrected QT (QTc) interval corrected for heart rate using Fridericia's formula (QTcF) > 450 msec for males and > 470 msec for females on the screening electrocardiogram (ECG).
    * Angina pectoris that requires the use of anti-anginal medication.
    * Ventricular arrhythmias except for benign premature ventricular contractions.
    * Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication.
    * Conduction abnormality requiring a pacemaker.
    * Valvular disease with documented compromise in cardiac function.
    * Symptomatic pericarditis.
12. Use of other investigational drugs within 30 days or 5 half-lives of initiation of study medication, whichever is longer.
13. Patients who are receiving treatment with medications known to be moderate and strong inhibitors or inducers of cytochrome P450 (CYP)isoenzyme 3A4/5 (CYP3A4) or drugs metabolized by CYP isoenzyme 2B6 (CYP2B6) or CYP isoenzyme 2C9 (CYP2C9) that have narrow therapeutic index, and that cannot be discontinued before starting treatment with LDE225. Medications that are strong CYP3A4/5 inhibitors should be discontinued at least 7 days and strong CYP3A4/5 inducers for at least 2 weeks prior to starting treatment with LDE225.
14. Patients are excluded if the use of warfarin (substrate of CYP2C9) is necessary and cannot be substituted since LDE225 is competitive inhibitor of CYP2C9 based on in vitro data.
15. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin laboratory test (> 5 milli-International Unit (mIU)/mL).
16. Patients who are not willing to apply highly effective contraception during the study and through the duration as defined below after the final dose of study treatment.

    Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, must use highly effective contraception during the study and through 6 months after the final dose of study treatment. Highly effective contraception is defined as either:
    * Total abstinence: When this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (i.e., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
    * Sterilization: Patient has had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
    * Male partner sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). [For female study patients, the vasectomised male partner should be the sole partner for that patient].
    * Use a combination of the following (both a+b):

      * Placement of a non-hormonal intrauterine device (IUD) or non-hormonal intrauterine system (IUS).
      * Barrier method of contraception: Condom or Occlusive cap (diaphragm or cervical vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.

    Note: Hormonal contraception methods (i.e. oral, injected, implanted) are not allowed as it cannot be ruled out that the study drug decreases the effectiveness of hormonal contraception.

    Note: Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (i.e. age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum follicle stimulating hormone (FSH) levels > 40 mIU/mL and estradiol < 20 pg/mL or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.

    Male patient must use highly effective (double barrier) methods of contraception (i.e., spermicidal gel plus condom) for the entire duration of the study, and continuing using contraception and refrain from fathering a child for 6 months following the study drug. A condom is required to be used also by vasectomized men in order to prevent delivery of the study treatment via seminal fluid.
17. Known human immunodeficiency virus (HIV) positivity.
18. Patients unwilling or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-02-10 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Safety of the combination assessed by evaluation of hematological and non-hematological toxicities at day 28 of cycle 1 | 1 month

SECONDARY OUTCOMES:
Clinical efficacy assessed by total percentage of responses, including all patients achieving CR, PR, marrow CR or hematologic improvement, evaluated according to IWG 2006 criteria after 6 treatment cycles | 6 months

OTHER OUTCOMES:
Overall survival | 3 years
  Overall survival measured from the date of enrollment to death or the date of last contact

CONTACTS AND LOCATIONS:
Overall Officials: Thomas PREBET, MD, Principal Investigator — Paoli Calmettes institute; Pierre FENAUX, MD, PHD, Study Director — Saint-Louis Hospital, Paris, France
Locations (24):
- France (24):
  - CHU d'Amiens, Amiens
  - CHU d'Angers, Angers
  - CH Henri Duffaut, Avignon
  - CH de la Côte Basque, Bayonne
  - Hôpital Avicenne, Bobigny
  - Hôpital Henri Mondor, Créteil
  - CHU de Grenoble, Grenoble
  - CH Le Mans, Le Mans
  - IPC-Unité d'Hématologie 3, Marseille
  - Centre Hospitalier de Meaux, Meaux
  - CHU de Montpellier, Montpellier
  - Hôpital Hôtel Dieu, Nantes
  - Centre Antoine Lacassagne, Nice
  - Hôpital Archet 1, Nice
  - CHU de Nîmes, Nîmes
  - Hôpital Saint Louis - Service Hématologie Sénior, Paris
  - Hôpital Saint-Louis - Service d'hématologie AJA, Paris
  - Hôpital Cochin, Paris
  - CHU de Haut-Lévèque, Pessac
  - CH Lyon Sud, Pierre-Bénite
  - CH Annecy Genevois, Pringy
  - Hôpital Henri Becquerel, Rouen
  - IUC Oncopole - Médecine interne, Toulouse
  - CHU Nancy-Brabois, Vandœuvre-lès-Nancy